CLINICAL TRIAL: NCT01469741
Title: Rehabilitation of Everyday Memory Impairment in Parkinson Disease: A Pilot Study
Acronym: REMI-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Erin Foster, Assistant Professor of Occupational Therapy, Neurology and Psychiatry, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201103176
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Prospective Memory Strategy — Prospective memory is central to performance in everyday life as it serves to bind together goal-directed actions and enables people to carry out their plans and wishes meaningfully and appropriately. Everyday prospective memory tasks include remembering to run errands, keep appointments, and turn off the stove after using it.

SUMMARY:
Cognitive impairment is common among non-demented individuals with Parkinson disease (PD) and is a significant source of disability and reduced quality of life. Unfortunately, there are no successful interventions to address these impairments. Prospective memory impairment is a particularly functionally- and clinically-relevant problem in PD. The investigator's project will determine if a targeted intervention strategy improves PD participants' prospective memory. The investigator's goal is to improve PD patients' everyday prospective memory so they can successfully perform desired activities and roles.

DETAILED DESCRIPTION:
Cognitive impairment is common among non-demented individuals with Parkinson disease (PD) and is a significant source of disability and reduced quality of life. Unfortunately, there are no successful interventions to address these impairments. Prospective memory impairment is a particularly functionally- and clinically-relevant problem in PD. The investigator's project will determine if a targeted intervention strategy improves PD participants' prospective memory. The investigator will use a randomized controlled design and a laboratory-based assessment of prospective memory to test the effect of the strategy in a controlled environment. The investigator will also see if PD participants, with support from an occupational therapist (OT), can generalize the strategy to their complex, real-world environments and tasks. Our goal is to improve PD patients' everyday prospective memory so they can successfully perform desired activities and roles.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be males and females over age 50 who meet criteria for idiopathic typical PD, are Hoehn & Yahr39 stage I-III (mild-moderate disease) and are treated with levodopa/carbidopa.

Exclusion Criteria:

* Possible dementia,
* treatment with certain medications that interfere with cognition (e.g., anticholinergics),
* change in medications over the study period, other neurological disorders, brain surgery (e.g., STN DBS),
* history of psychotic disorder or significant current psychiatric disorder, or any condition that would interfere with testing (e.g., vision problems).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Foster, OTD, OTR/L, Principal Investigator — Washington University School of Medicine, Department of Occupational Therapy
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States